CLINICAL TRIAL: NCT00983437
Title: A 12-Month, Open-Label Study to Evaluate the Safety, Tolerability, and Efficacy of Armodafinil (150 and 250 mg/Day) as Treatment for Patients With Excessive Sleepiness Associated With Mild or Moderate Closed Traumatic Brain Injury
Brief Title: Study to Evaluate the Safety, Tolerability, and Efficacy of Armodafinil as Treatment for Patients With Excessive Sleepiness Associated With Mild or Moderate Closed Traumatic Brain Injury
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study has been stopped by sponsor decision
Sponsor: Cephalon, Inc. (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C10953/3069/ES/MN
Record Dates: First submitted 2009-09-09; First posted 2009-09-24 (Estimated); Results first posted 2013-10-18 (Estimated); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Modafinil

ARMS (1):
- Armodafinil (Experimental): Armodafinil tablets 150 mg or 250 mg administered orally, once daily in the morning.
  Interventions: Drug: Armodafinil

INTERVENTIONS:
Drug: Armodafinil
  Other Names: CEP-10953

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of long-term (12 months) armodafinil treatment in patients with excessive sleepiness associated with mild or moderate closed traumatic brain injury (TBI).

ELIGIBILITY:
Patients enrolled in this study will be rollover patients (those who completed the previous double-blind efficacy study C10953/3067/ES/MN) and new patients (those who did not participate in the C10953/3067/ES/MN study).

Inclusion Criteria (for New Patients):

* The patient has a mild (Glasgow Coma Scale [GCS] score = 13-15) or moderate (GCS score = 9-12) closed traumatic brain injury (TBI) at the time of the injury, and the injury occurred 1 to 10 years prior to screening.
* The patient has a Glasgow Outcome Scale score of 5.
* The patient has an Epworth Sleepiness Scale (ESS) score of at least 10.
* The patient has a mean sleep latency on the Multiple Sleep Latency Test (MSLT) (average of 4 naps) of less than 8 minutes.
* The patient has a Clinical Global Impression of Severity of Illness (CGI-S) rating relating to their excessive sleepiness of 4 or more.
* The patient has a complaint of excessive sleepiness (at least 5 days/week on average) for at least 3 months, and the excessive sleepiness began within 12 months of the TBI identified according to the first inclusion criterion.
* Written informed consent was obtained.
* If admitted to an in-patient treatment facility, the patient was discharged at least 1 month prior to the screening visit.
* The patient does not have any medical or psychiatric disorders that could account for the excessive sleepiness.
* Women of childbearing potential (not surgically sterile or 2 years postmenopausal), used a medically accepted method of contraception, and continued use of 1 of those methods for the duration of the study (and for 30 days after participation in the study).
* The patient is in otherwise good health, as judged by the investigator, on the basis of a medical and psychiatric history, physical examination, electrocardiogram (ECG), serum chemistry, hematology, and urinalysis.
* The patient is willing and able to comply with study restrictions and attend regularly scheduled clinic visits as specified in the protocol.
* The patient has an mini-mental state examination (MMSE) score of more than 26 at the screening visit.
* The patient was on stable dosages of medications (allowed by the protocol) for a minimum of 3 months (selective serotonin reuptake inhibitor [SSRIs] and serotonin and norepinephrine reuptake inhibitor [SNRIs]), 8 weeks (contraceptives), or 4 weeks (all other allowed medication) before the screening visit and is not likely to require a change in therapy for at least 12 weeks on the basis of the investigators' assessment.
* The patient has no other head injuries that, based on medical record documentation or history from the patient and reliable informant (if available), were temporally related to the onset or to any worsening of excessive sleepiness.
* The patient has no other head injury fulfilling the criteria for TBI within ±1 year of the TBI identified according to the first inclusion criterion.
* The patient has a habitual bedtime between 2100 and 2400.

Inclusion Criteria (for Rollover Patients from Study C10953/3067/ES/MN):

* The patient has completed 12 weeks of double-blind treatment in Study C10953/3067/ES/MN.
* Written informed consent was obtained.
* Women of childbearing potential (not surgically sterile or 2 years postmenopausal), used a medically accepted method of contraception and agreed to continue use 1 of those methods for the duration of the study and for 30 days after participation in the study.
* The patient is in otherwise good health, as judged by the investigator, on the basis of a medical and psychiatric history, physical examination, ECG, serum chemistry, hematology, and urinalysis.
* The patient is willing and able to comply with study restrictions and to remain at the clinic for the required duration during the study period, and was willing to return to the clinic for the follow-up evaluation as specified in the protocol.

Exclusion Criteria (for New Patients):

* The patient has a history of 2 or more episodes of transient loss of consciousness without clear medical explanation, or has a history of known or suspected pseudo seizure (psychogenic seizure). Patients with a history of seizure or epilepsy may be eligible following discussion with the medical monitor.
* The patient requires, or is likely to require, treatment with anticonvulsant medication during the study; or has taken anticonvulsant medication within 6 months before the screening visit.
* The patient has an unstable or uncontrolled medical (including illnesses related to the cardiovascular, renal, or hepatic systems) or surgical condition (treated or untreated) or was not a suitable candidate for treatment with armodafinil, as judged by the investigator.
* The patient has had neurosurgery involving the brain or brainstem.
* The patient has a history of schizophrenia, bipolar disorder, psychotic depression, or other psychotic episode.
* The patient has any current Axis I disorder (including depression and posttraumatic stress disorder [PTSD]), as assessed by Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (SCID). Patients with any Axis II disorder, that in the opinion of the investigator, would affect patient participation in the study or full compliance with study procedures.
* The patient has a history of, or currently meets The International Classification of Sleep Disorders, Edition 2 (ICSD-2) criteria for any other sleep disorder associated with excessive daytime sleepiness; or the patient has a history of idiopathic hypersomnia, insomnia (requiring treatment), or sleep disorder before the development of the TBI.
* The patient has 85% or less sleep efficiency (sleep duration ÷ time in bed x 100%) as determined from Nocturnal Polysomnography (NPSG).
* The patient has any disorder that may have interfered with drug absorption, distribution, metabolism, or excretion.
* The patient has used any medications including over-the-counter (OTC) medicines disallowed by the protocol within 7 days or 5 half-lives (medication or its active metabolites), whichever is longer.
* The patient has a need for chronic pain medications.
* In the judgment of the investigator, the patient has a clinically significant deviation from normal in the physical examination.
* In the judgment of the investigator, the patient has any clinically significant ECG finding.
* The patient has a diagnosis of any type of dementia.
* The patient has a history of suicidal ideation (considered by the investigator to be of clinical significance), or is suicidal.
* The patient has a known hypersensitivity to armodafinil, racemic modafinil, or any component of the study drug tablets. Armodafinil tablets contained the following inactive ingredients: croscarmellose sodium, lactose, magnesium stearate, microcrystalline cellulose, povidone, and pregelatinized starch.
* The patient has a history of any clinically significant cutaneous drug reaction, or a history of clinically significant hypersensitivity reaction, including multiple allergies or drug reactions.
* The patient has a clinical laboratory test value(s) outside the range(s) specified in the protocol (or any other clinically significant laboratory abnormality), and the medical monitor had not provided written approval for study participation.
* The subject has a history (within the past 5 years) of alcohol, narcotic, or any other drug abuse (with the exception of nicotine) as defined by the Diagnostic and Statistical Manual of Mental Disorders of the American Psychiatric Association, 4th Edition (DSM-IV-TR) or the patient had current evidence of substance use, without medical explanation, confirmed by results of a urine drug screen (UDS).
* The patient has taken armodafinil, modafinil, or other stimulant medication for excessive sleepiness within 1 month of the screening visit.
* The patient is a pregnant or lactating woman.
* The patient is known to have tested positive for human immunodeficiency virus (HIV).
* The patient consumes an average of more than 600 mg of caffeine per day, including coffee, tea and/or other caffeine-containing beverages or food.
* The patient has used any investigational drug within 1 month before the screening visit.
* The patient is receiving workmen's compensation or was in active litigation with regard to TBI.
* The patient has a Self-Reported Hamilton Depression Rating Scale, 6 Item Version (S-HAM-D6) score of more than 4.

Exclusion Criteria (for Rollover Patients from Study C10953/3067/ES/MN):

* The patient has any clinically significant unstable or uncontrolled medical, surgical, or psychiatric conditions (treated or untreated) or may not be a suitable candidate for treatment with armodafinil, as judged by the investigator or medical monitor.
* The patient has current evidence of active psychosis, including stimulant-induced psychosis or mania.
* The patient has current evidence of non-medical substance use confirmed by results of a UDS.
* The patient has used any medications including OTC medicines disallowed by the protocol (except armodafinil use in study 3067) within 7 days or 5 half-lives of the drug and its active metabolites, whichever is longer.
* The patient has a clinically significant deviation from normal in the physical examination as judged by the investigator.
* The patient has a clinically significant laboratory abnormality, as judged by the investigator, without prior written approval by the medical monitor.
* The patient has hypersensitivity to armodafinil or modafinil, or any of the excipients of either.
* The patient is a pregnant or lactating woman.
* The patient is unlikely to comply with the study protocol, or is unsuitable for any other reason, as judged by the investigator.
* The patient consumes an average of more than 600 mg of caffeine per day (approximately equivalent to 5 or more cups of coffee), including coffee, tea, and/or other caffeine-containing beverages or food.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2009-08-31 (Actual); Primary Completion 2011-01-31 (Actual); Study Completion 2011-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor's Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (61):
- United States (61):
  - Teva Investigational Site 58, Birmingham, Alabama
  - Teva Investigational Site 62, Tucson, Arizona
  - Teva Investigational Site 16, Hot Springs, Arkansas
  - Teva Investigational Site 5, Little Rock, Arkansas
  - Teva Investigational Site 44, Fountain Valley, California
  - Teva Investigational Site 49, La Palma, California
  - Teva Investigational Site 51, La Palma, California
  - Teva Investigational Site 55, San Diego, California
  - Teva Investigational Site 33, San Diego, California
  - Teva Investigational Site 53, Santa Monica, California
  - Teva Investigational Site 69, Wallingford, Connecticut
  - Teva Investigational Site 52, Hallandale, Florida
  - Teva Investigational Site 47, Miami, Florida
  - Teva Investigational Site 1, Orlando, Florida
  - Teva Investigational Site 18, Pembroke Pines, Florida
  - Teva Investigational Site 10, Spring Hill, Florida
  - Teva Investigational Site 38, St. Petersburg, Florida
  - Teva Investigational Site 17, Tampa, Florida
  - Teva Investigational Site 12, Atlanta, Georgia
  - Teva Investigational Site 14, Atlanta, Georgia
  - Teva Investigational Site 68, Gainesville, Georgia
  - Teva Investigational Site 67, Macon, Georgia
  - Teva Investigational Site 15, Suwanee, Georgia
  - Teva Investigational Site 46, Chicago, Illinois
  - Teva Investigational Site 54, Chicago, Illinois
  - Teva Investigational Site 59, Chicago, Illinois
  - Teva Investigational Site 28, Danville, Indiana
  - Teva Investigational Site 19, Fort Wayne, Indiana
  - Teva Investigational Site 2, Indianapolis, Indiana
  - Teva Investigational Site 39, Indianapolis, Indiana
  - Teva Investigational Site 41, Iowa City, Iowa
  - Teva Investigational Site 9, Shawnee Mission, Kansas
  - Teva Investigational Site 48, Louisville, Kentucky
  - Teva Investigational Site 32, Chevy Chase, Maryland
  - Teva Investigational Site 37, Belmont, Massachusetts
  - Teva Investigational Site 22, Saginaw, Michigan
  - Teva Investigational Site 7, Hattiesburg, Mississippi
  - Teva Investigational Site 42, St Louis, Missouri
  - Teva Investigational Site 56, Lincoln, Nebraska
  - Teva Investigational Site 63, New York, New York
  - Teva Investigational Site 36, West Seneca, New York
  - Teva Investigational Site 11, Durham, North Carolina
  - Teva Investigational Site 45, Winston-Salem, North Carolina
  - Teva Investigational Site 31, Cincinnati, Ohio
  - Teva Investigational Site 34, Cincinnati, Ohio
  - Teva Investigational Site 57, Middleburg Heights, Ohio
  - Teva Investigational Site 30, Toledo, Ohio
  - Teva Investigational Site 3, Oklahoma City, Oklahoma
  - Teva Investigational Site 64, Clarks Summit, Pennsylvania
  - Teva Investigational Site 13, Jefferson Hills, Pennsylvania
  - Teva Investigational Site 65, Columbia, South Carolina
  - Teva Investigational Site 61, Germantown, Tennessee
  - Teva Investigational Site 60, Austin, Texas
  - Teva Investigational Site 25, Dallas, Texas
  - Teva Investigational Site 8, Houston, Texas
  - Teva Investigational Site 20, Houston, Texas
  - Teva Investigational Site 23, San Antonio, Texas
  - Teva Investigational Site 35, Midvale, Utah
  - Teva Investigational Site 66, Midvale, Utah
  - Teva Investigational Site 24, Richmond, Virginia
  - Teva Investigational Site 50, West Allis, Wisconsin

REFERENCES:
- [Derived] Menn SJ, Yang R, Lankford A. Armodafinil for the treatment of excessive sleepiness associated with mild or moderate closed traumatic brain injury: a 12-week, randomized, double-blind study followed by a 12-month open-label extension. J Clin Sleep Med. 2014 Nov 15;10(11):1181-91. doi: 10.5664/jcsm.4196. PMID 25325609

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of patients with excessive sleepiness associated with mild or moderate traumatic brain injury (TBI) who had completed study C10953/3067/ES/MN (NCT00893789) and were considered to be eligible for enrollment into the current study, 49 patients at 25 centers in the United States were enrolled. No new patients were screened for the study.
Pre-assignment Details: Of 49 participants enrolled, 2 were withdrawn before taking any study drug for reasons of protocol violation and noncompliance with study procedures, respectively.
Period: Overall Study
Arm/Group | Armodafinil
Started | 47
Safety Analysis Set (SAS) | 47 (Participants who received at least 1 dose of study drug were evaluable for safety.)
Full Analysis Set (FAS) | 45 (Participants had to have at least 1 postbaseline efficacy assessment to be evaluable for efficacy.)
Completed | 0 (Completed 12 months of treatment with armodafinil.)
Not Completed | 47
Not completed — Adverse Event | 9
Not completed — Lack of Efficacy | 1
Not completed — Withdrawal by Subject | 8
Not completed — Noncompliance to Study Procedures | 1
Not completed — Lost to Follow-up | 2
Not completed — Other Reason | 26

BASELINE CHARACTERISTICS:
Population: Baseline Analysis Population includes 2 participants who were enrolled but not treated.
Arm/Group | Armodafinil
Number analyzed (Participants) | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.1 (10.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 30
Race/Ethnicity, Customized [Number; unit: participants]
  White | 43
  Black | 3
  Asian | 2
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), Deaths and Discontinuations Due to AEs
Description: AE=any untoward medical occurrence that develops or worsens in severity during the conduct of the clinical study of a pharmaceutical product and does not necessarily have a causal relationship to the study drug. SAE=any AE that resulted in any of the following: death; a life-threatening adverse event; inpatient hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity; a congenital anomaly or birth defect; an important medical event that required medical intervention to prevent 1 of the outcomes listed in this definition. Treatment-related AEs=definite, probable, possible, or missing relationship to study drug. Protocol-defined AEs=treatment-emergent adverse events associated with skin rash, hypersensitivity reaction, emergent suicidal ideation or suicide attempt, depression, psychosis, and seizure or suspected seizure were considered to be of potential clinical importance. DB=double-blind portion of the study (NCT00893789).
Time Frame: Assessed from Screening through end of treatment; median (full range) of treatment was 98 (5.0 to 326.0) days.
Population: Safety Analysis Set (study participants who received at least 1 dose of study drug)
Measure: Number; unit: participants
Arm/Group | Armodafinil
Number analyzed (Participants) | 47
participants
  Any AE | 29
  Severe AEs | 0
  Treatment-related AEs | 17
  Deaths | 0
  SAEs (Other Than Deaths) | 1
  Discontinuations (DCs) Due to AEs | 7
  Protocol-defined AEs | 3
  DCs due to AEs with onset during DB phase | 2

2. Primary Outcome: Safety and Tolerability: Concomitant Medication Usage In Participants Throughout the Study
Description: Therapeutic classification of concomitant medications used by participants throughout the study. Participants are counted only once in each therapeutic class category.
Time Frame: Assessed from Screening through end of treatment; median (full range) of treatment was 98 (5.0 to 326.0) days.
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | Armodafinil
Number analyzed (Participants) | 47
participants
  Participants receiving any concomitant medication | 39
  All other therapeutic products | 1
  Analgesics | 10
  Anesthetics | 1
  Anti-anemic preparations | 1
  Antibacterials for systemic use | 4
  Anti-emetics and antinauseants | 1
  Antigout preparations | 1
  Antihistamines for systemic use | 4
  Anti-inflammatory and antirheumatic products | 16
  Antimycotics for systemic use | 1
  Antithrombotic agents | 1
  Beta blocking agents | 1
  Cardiac therapy | 1
  Corticosteroids for systemic use | 1
  Cough and cold preparations | 2
  Drugs for acid-related disorders | 3
  Drugs for obstructive airway diseases | 3
  Drugs used in diabetes | 1
  General nutrients | 1
  Lipid-modifying agents | 11
  Nasal preparations | 4
  Other gynecologicals | 2
  Psychoanaleptics | 1
  Psycholeptics | 2
  Sex hormones and modulators of the genital system | 7
  Thyroid therapy | 1
  Unspecified herbal | 4
  Vitamins | 12

3. Primary Outcome: Safety and Tolerability: Number of Participants With Clinically Significant Serum Chemistry Test Results
Description: Criteria for clinically significant abnormal serum chemistry values: alanine aminotransferase (ALT) ≥3x upper limit of normal (ULN); aspartate aminotransferase (AST) ≥3x ULN; alkaline phosphatase ≥3x ULN; gamma-glutamyl transpeptidase (GGT) ≥3x ULN; lactate dehydrogenase (LDH) ≥3x ULN; blood urea nitrogen (BUN) ≥10.71 mmol/L; creatinine ≥177 μmol/L; uric acid, men ≥625 μmol/L, women ≥506 μmol/L; bilirubin (total) ≥34.2 μmol/L.
Time Frame: Assessed at Screening, Months 6 and 12 (or last postbaseline observation); median (full range) of treatment was 98 (5.0 to 326.0) days.
Population: Participants in the Safety Analysis Set who had a baseline and at least one post-baseline value.
Measure: Number; unit: participants
Arm/Group | Armodafinil
Number analyzed (Participants) | 38
participants
  Participants with at least 1 abnormality (overall) | 3
  Blood Urea Nitrogen >=10.71 | 2
  Uric Acid >=625 (male) or >=506 (female) µmol/L | 1

4. Primary Outcome: Safety and Tolerability: Number of Participants With Clinically Significant Abnormal Vital Signs Measurements
Description: Criteria for clinically significant abnormal vital signs values: pulse, ≥120 beats per minute (bpm) and increase from baseline of ≥15 bpm or ≤50 bpm and decrease from baseline of ≥15 bpm; systolic blood pressure, ≥180 mm Hg and increase from baseline of ≥20 mm Hg or ≤90 mm Hg and decrease from baseline of ≥20 mm Hg; diastolic blood pressure, ≥105 mm Hg and increase from baseline of ≥15 mm Hg or ≤50 mm Hg and decrease from baseline of ≥15 mm Hg; temperature >38.3º celsius (C) and change from baseline of ≥1.1°C. Baseline was defined as the baseline value from the double-blind study C10953/3067/ES/MN (NCT00893789) from which the participants entered into this open-label study.
Time Frame: Baseline, Week 2, Months 1, 2, 3, 6, 9, and 12 (or last postbaseline observation); median (full range) of treatment was 98 (5.0 to 326.0) days.
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | Armodafinil
Number analyzed (Participants) | 47
participants | 0

5. Secondary Outcome: Change From Baseline in Epworth Sleepiness Scale (ESS) at Week 2 and Months 1, 2, 3, 6, 9, and Endpoint (Month 12 or Last Postbaseline Observation)
Description: The participant's evaluation of excessive daytime sleepiness was measured by the ESS. The ESS score is based on responses to questions referring to 8 everyday situations (eg, sitting and reading, talking to someone, being stopped in traffic) and reflects a patient's propensity to fall asleep in those situations. The ESS score is derived from the sum of the values from questions corresponding to the 8 situations. Scores for the ESS range from 0 to 24, with a higher score indicating a greater daytime sleepiness. This test was self-administered. Baseline was defined as the baseline value from the double-blind study C10953/3067/ES/MN (NCT00893789) from which the participants entered into this open-label study.
Time Frame: Baseline, Week 2 and Months 1, 2, 3, 6, 9, and Endpoint (Month 12 or last postbaseline observation); median (full range) of treatment was 98 (5.0 to 326.0) days.
Population: Full Analysis Set = participants in the Safety Analysis Set who had at least 1 post-baseline efficacy assessment; n=number of participants with value at baseline and given time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Armodafinil
Number analyzed (Participants) | 45
units on a scale
  Baseline (BL; n=45) | 14.8 (2.60)
  Change from BL at Week 2 (n=41) | -8.0 (4.42)
  Change from BL at Month 1 (n=35) | -8.5 (4.37)
  Change from BL at Month 2 (n=30) | -9.0 (3.56)
  Change from BL at Month 3 (n=22) | -9.0 (3.53)
  Change from BL at Month 6 (n=11) | -10.0 (3.26)
  Change from BL at Month 9 (n=4) | -10.3 (4.79)
  Change from BL at Endpoint (n=45) | -9.0 (4.48)

6. Secondary Outcome: Change From Baseline in Clinical Global Impression of Severity of Illness (CGI-S) at Week 2 and Months 1, 2, 3, 6, 9, and Endpoint (Month 12 or Last Postbaseline Observation)
Description: The clinician's rating of disease severity as assessed by the Clinical Global Impression of Severity (CGI-S). CGI-S assesses the severity of the subject's condition on a 7-point scale ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill); the 7 categories include the following: normal-shows no sign of illness, borderline ill, mildly (slightly) ill, moderately ill, markedly ill, severely ill, and among the most extremely ill. Baseline was defined as the baseline value from the double-blind study C10953/3067/ES/MN (NCT00893789) from which the participants entered into this open-label study.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Armodafinil
Number analyzed (Participants) | 45
units on a scale
  Baseline (BL; n=45) | 4.4 (0.53)
  Change from BL at Week 2 (n=41) | -1.9 (1.04)
  Change from BL at Month 1 (n=35) | -2.1 (1.09)
  Change from BL at Month 2 (n=30) | -2.6 (0.81)
  Change from BL at Month 3 (n=22) | -2.4 (0.73)
  Change from BL at Month 6 (n=11) | -2.5 (1.29)
  Change from BL at Month 9 (n=4) | -3.3 (0.96)
  Change from BL at Endpoint (n=45) | -2.2 (1.15)

7. Secondary Outcome: Percentage of Participants With Improvement on the Clinical Global Impression of Severity of Illness (CGI-S) at Week 2 and Months 1, 2, 3, 6, 9, and Endpoint (Month 12 or Last Postbaseline Observation)
Description: The clinician's rating of disease severity as assessed by the Clinical Global Impression of Severity (CGI-S). CGI-S assesses the severity of the subject's condition on a 7-point scale ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill); the 7 categories include the following: normal-shows no sign of illness, borderline ill, mildly (slightly) ill, moderately ill, markedly ill, severely ill, and among the most extremely ill. Improvement is defined as at least 1 point improvement from baseline. Baseline was defined as the baseline value from the double-blind study C10953/3067/ES/MN (NCT00893789) from which the participants entered into this open-label study.
Time Frame: Week 2 and Months 1, 2, 3, 6, 9, and Endpoint (Month 12 or last postbaseline observation); median (full range) of treatment was 98 (5.0 to 326.0) days.
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Armodafinil
Number analyzed (Participants) | 45
percentage of participants
  Improved at Week 2 (n=41) | 95
  Not Improved at Week 2 (n=41) | 5
  Improved at Month 1 (n=35) | 97
  Not Improved at Month 1 (n=35) | 3
  Improved at Month 2 (n=30) | 100
  Not Improved at Month 2 (n=30) | 0
  Improved at Month 3 (n=22) | 100
  Not Improved at Month 3 (n=22) | 0
  Improved at Month 6 (n=11) | 91
  Not Improved at Month 6 (n=11) | 9
  Improved at Month 9 (n=4) | 100
  Not Improved at Month 9 (n=4) | 0
  Improved at Endpoint (n=45) | 93
  Not Improved at Endpoint (n=45) | 7

8. Secondary Outcome: Change From Baseline in Traumatic Brain Injury - Work Instability Scale (TBI-WIS) Score Values at Months 3, 6, 9, and Endpoint (Month 12 or Last Postbaseline Observation)
Description: The TBI-WIS is a validated participant-rated instrument for assessing a participant's functional ability after TBI and the functional demands of their job. The assessment consists of 36 questions to which the participant responded with a "true" or "not true" answer. To score the questionnaire, the number of "true" responses is counted: if < 2, the risk for work instability is low; 2 to 23, the risk is medium; and >23, the risk is high. Score range is 0 (lowest risk for work instability) to 36 (highest risk for work instability). Baseline was defined as the baseline value from the double-blind study C10953/3067/ES/MN (NCT00893789) from which the participants entered into this open-label study.
Time Frame: Baseline, Months 3, 6, 9, and Endpoint (Month 12 or last postbaseline observation); median (full range) of treatment was 98 (5.0 to 326.0) days.
Population: Participants in the Full Analysis Set (those in the Safety Analysis Set with at least 1 post-baseline efficacy assessment) with a TBI-WIS score at baseline; n=number of participants with value at baseline and given time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Armodafinil
Number analyzed (Participants) | 34
units on a scale
  Baseline (BL; n=34) | 9.6 (6.93)
  Change from BL at Month 3 (n=19) | -3.1 (5.87)
  Change from BL at Month 6 (n=10) | -2.5 (7.32)
  Change from BL at Month 9 (n=3) | -7.3 (2.52)
  Change from BL at Endpoint (n=34) | -4.6 (6.52)

9. Primary Outcome: Safety and Tolerability: Number of Participants With Clinically Significant Abnormal Hematology Test Results
Description: Criteria for clinically significant abnormal hematology values: hematocrit, men <0.37 L/L or women <0.32 L/L; hemoglobin, men ≤115 g/L or women ≤95 g/L; white blood cell (WBC) count ≤3x10^9/L or ≥20x10^9/L; eosinophils ≥10%; absolute neutrophil count (ANC) ≤1x10^9/L; platelet count ≤75x10^9/L or ≥700x10^9/L.
Time Frame: as for outcome 3
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | Armodafinil
Number analyzed (Participants) | 47
participants | 0

10. Primary Outcome: Safety and Tolerability: Number of Participants With Clinically Significant Abnormal Urinalysis Results
Description: Criteria for clinically significant abnormal urinalysis values: blood (hemoglobin) ≥2 unit increase from baseline; glucose ≥2 unit increase from baseline; ketones ≥2 unit increase from baseline; total protein ≥2 unit increase from baseline. Baseline was defined as the baseline value from the double-blind study C10953/3067/ES/MN (NCT00893789) from which the participants entered into this open-label study.
Time Frame: Baseline, Months 6 and 12 (or last postbaseline observation); median (full range) of treatment was 98 (5.0 to 326.0) days.
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | Armodafinil
Number analyzed (Participants) | 47
participants | 0

11. Primary Outcome: Safety and Tolerability: Number of Participants With Notable Blood Pressure Values Per World Health Organization Criteria
Description: Criteria for World Health Organization (WHO) notable blood pressure (BP) values: systolic blood pressure ≥140 mm Hg plus increase of ≥10% from baseline; diastolic blood pressure ≥90 mm Hg plus increase of ≥10% from baseline. Baseline was defined as the baseline value from the double-blind study C10953/3067/ES/MN (NCT00893789) from which the participants entered into this open-label study.
Time Frame: as for outcome 4
Population: Safety Analysis Set; participants with a baseline and postbaseline value.
Measure: Number; unit: participants
Arm/Group | Armodafinil
Number analyzed (Participants) | 45
participants
  Participants with at least 1 notable BP value | 6
  Sitting systolic BP >=140 mm Hg + Increase >=10% | 4
  Sitting diastolic BP >=90 mm Hg + Increase >=10% | 3

12. Primary Outcome: Safety and Tolerability: Electrocardiogram (ECG) Findings Shifts From Baseline to Overall
Description: Number of participants with shifts from normal/abnormal 12-lead ECG findings at baseline (BL) to (→) normal/abnormal findings overall are presented. For overall, the worst postbaseline finding (the abnormal finding if there are both normal and abnormal findings) for the participant between baseline and endpoint (defined as last postbaseline observation, up to Week 12) is summarized. Any ECG finding that was judged by the investigator as a clinically meaningful change (worsening) compared to baseline was recorded as an adverse event. Baseline was defined as the baseline value from the double-blind study C10953/3067/ES/MN (NCT00893789) from which the participants entered into this open-label study.
Time Frame: Baseline through Endpoint (Month 12 or last postbaseline observation); median (full range) of treatment was 98 (5.0 to 326.0) days.
Population: Safety Analysis Set; only those participants with both baseline and endpoint ECG findings are summarized.
Measure: Number; unit: participants
Arm/Group | Armodafinil
Number analyzed (Participants) | 35
participants
  Normal at BL → Normal Overall | 17
  Normal at BL→ Abnormal Overall | 4
  Abnormal at BL→ Normal Overall | 3
  Abnormal at BL → Abnormal Overall | 11

13. Primary Outcome: Safety and Tolerability: Physical Examination Findings Shifts From Baseline to Endpoint (Month 12 or Last Postbaseline Observation)
Description: Number of participants with shifts from normal/abnormal physical examination findings at baseline (BL) to (→) normal/abnormal findings at endpoint (EP). Shifts (normal and abnormal) from baseline to endpoint are summarized using participant counts for each physical examination category. A newly diagnosed finding was defined as being normal or missing at baseline and abnormal at least once during the study. Any physical examination finding that was judged by the investigator as a clinically significant change (worsening) compared to a baseline value was considered an adverse event. HEENT= head, eyes, ears, nose, throat. Baseline was defined as the baseline value from the double-blind study C10953/3067/ES/MN (NCT00893789) from which the participants entered into this open-label study.
Time Frame: as for outcome 12
Population: Safety Analysis Set; only those participants with both baseline and endpoint physical examination findings are summarized.
Measure: Number; unit: participants
Arm/Group | Armodafinil
Number analyzed (Participants) | 39
participants
  General Appearance: Normal at BL→Normal at EP | 37
  General Appearance: Normal at BL→ Abnormal at EP | 2
  General Appearance: Abnormal at BL→ Normal at EP | 0
  General Appearance: Abnormal at BL→Abnormal at EP | 0
  HEENT: Normal at BL→Normal at EP | 37
  HEENT: Normal at BL→Abnormal at EP | 1
  HEENT: Abnormal at BL→Normal at EP | 1
  HEENT: Abnormal at BL→Abnormal at EP | 0
  Chest/Lungs: Normal at BL→Normal at EP | 39
  Chest/Lungs: Normal at BL→Abnormal at EP | 0
  Chest/Lungs: Abnormal at BL→Normal at EP | 0
  Chest/Lungs: Abnormal at BL→Abnormal at EP | 0
  Heart: Normal at BL→Normal at EP | 38
  Heart: Normal at BL→Abnormal at EP | 1
  Heart: Abnormal at BL→Normal at EP | 0
  Heart: Abnormal at BL→Abnormal at EP | 0
  Abdomen: Normal at BL→Normal at EP | 38
  Abdomen: Normal at BL→Abnormal at EP | 1
  Abdomen: Abnormal at BL→Normal at EP | 0
  Abdomen: Abnormal at BL→Abnormal at EP | 0
  Musculoskeletal: Normal at BL→Normal at EP | 38
  Musculoskeletal: Normal at BL→Abnormal at EP | 1
  Musculoskeletal: Abnormal at BL→Normal at EP | 0
  Musculoskeletal: Abnormal at BL→Abnormal at EP | 0
  Skin: Normal at BL→Normal at EP | 35
  Skin: Normal at BL→Abnormal at EP | 0
  Skin: Abnormal at BL→Normal at EP | 0
  Skin: Abnormal at BL→Abnormal at EP | 4
  Lymph Nodes: Normal at BL→Normal at EP | 34
  Lymph Nodes: Normal at BL→Abnormal at EP | 0
  Lymph Nodes: Abnormal at BL→Normal at EP | 1
  Lymph Nodes: Abnormal at BL→Abnormal at EP | 0
  Neurological: Normal at BL→Normal at EP | 37
  Neurological: Normal at BL→Abnormal at EP | 1
  Neurological: Abnormal at BL→Normal at EP | 1
  Neurological: Abnormal at BL→Abnormal at EP | 0

14. Primary Outcome: Number of Participants Answering "Yes" to Any Question on the Columbia-Suicide Severity Rating Scale Since Last Visit Version (C-SSRS SLV) at Week 2, Months 1, 2, 3, 6, 9, and Endpoint (Month 12, or Last Postbaseline Observation)
Description: The percentage of participants answering 'yes' to any of the 9 yes/no questions about suicidal behaviors, ideations, and acts at given time points are presented. The C-SSRS captures occurrence, severity, and frequency of suicide-related thoughts and behaviors since last visit (SLV). Questions included the presence (yes) or absence (no) of the following: a wish to be dead; nonspecific active suicidal thoughts; actual suicide attempt; non-suicidal self-injurious behavior; interrupted attempt; aborted attempt; suicidal behavior; preparatory suicidal acts or behavior; and completed suicide.
Time Frame: Week 2, Months 1, 2, 3, 6, 9, and Endpoint (Month 12, or last postbaseline observation); median (full range) of treatment was 98 (5.0 to 326.0) days.
Population: Safety Analysis Set; n=number of participants with nonmissing value at given time point.
Measure: Number; unit: participants
Arm/Group | Armodafinil
Number analyzed (Participants) | 47
participants
  Week 2 (n=18), yes to any question | 0
  Month 1 (n=18), yes to any question | 0
  Month 2 (n=18), yes to any question | 0
  Month 3 (n=13), yes to any question | 0
  Month 6 (n=10), yes to any question | 0
  Month 9 (n=4), yes to any question | 0
  Endpoint (n=36), yes to 'Wish to Be Dead' question | 1
  Endpoint (n=36), yes to all other questions | 0

15. Primary Outcome: Change From Baseline in the Total Score From the Self-Reported Hamilton Depression Rating Scale, 6 Item Version (S-HAM-D6) at Week 2, Months 1, 2, 3, 6, 9, and Endpoint (Month 12, or Last Postbaseline Observation)
Description: The self-reported S-HAM-D6 is a validated scale developed from the core depressive items of the 17 Item Hamilton Depression Inventory (HAM-D17). The HAM-D6 (Items 1, 2, 7, 8, 10, 13 from the 17-item HAMD) evaluates "core" symptoms of Major Depressive Disorder (MDD). The assessment consists of 6 items representing depressed mood, guilt, work and activities, retardation, psychic anxiety, and general somatic symptoms. Each item is evaluated and scored using either a 5-point scale (e.g. absent, mild, moderate, severe, very severe) or a 3-point scale (e.g. absent, mild, marked). Total scores range from 0 (normal) to 22 (severe). Scores greater than 12 indicate moderate to severe depression. Baseline was defined as the baseline value from the double-blind study C10953/3067/ES/MN (NCT00893789) from which the participants entered into this open-label study.
Time Frame: Baseline, Week 2, Months 1, 2, 3, 6, 9, and Endpoint (Month 12, or last postbaseline observation); median (full range) of treatment was 98 (5.0 to 326.0) days.
Population: Participants in the Safety Analysis Set with a Baseline value; n=number of participants with baseline and postbaseline value at given time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Armodafinil
Number analyzed (Participants) | 13
units on a scale
  Baseline (BL; n=13) | 1.4 (1.33)
  Change from BL at Week 2 (n=13) | 0.9 (3.43)
  Change from BL at Month 1 (n=12) | 0.2 (2.41)
  Change from BL at Month 2 (n=9) | 0.0 (2.35)
  Change from BL at Month 3 (n=1) | -1.0 (NA) — Only 1 participant measured.
  Change from BL at Month 6 (n=0) | NA (NA) — No participants had available measurements at this time point.
  Change from BL at Month 9 (n=0) | NA (NA) — No participants had available measurements at this time point.
  Change from BL at Endpoint (n=13) | 0.0 (2.65)

16. Secondary Outcome: Change From Baseline in the Medical Outcomes Study 6-Item Cognitive Functioning Scale (MOS-CF6) Total Score at Months 3, 6, 9, and Endpoint (Month 12 or Last Postbaseline Observation)
Description: The MOS-CF 6 is an instrument to assess patient self-reported cognitive function. Items were selected to cover 6 relevant aspects of cognitive functioning as follows: confusion, concentration/thinking, attention, memory, reasoning, problem solving, and processing speed. The CF 6-item responses include 6 choices, ranging from "none of the time" to "all of the time." The CF-6 is scored by summing responses across the 6 items and converting the total to a 0- to 100-point scale, with higher scores indicating better cognitive functioning. Baseline was defined as the baseline value from the double-blind study C10953/3067/ES/MN (NCT00893789) from which the participants entered into this open-label study.
Time Frame: Baseline, Months 3, 6, 9, and 12 (or last postbaseline observation)
Population: Changes from baseline in MOS-CF6 total score were not summarized. This assessment was not performed in study C10953/3067/ES/MN (NCT00893789); therefore, the data obtained at screening for the current study would represent true baseline data only for new participants, of which there were none.
Arm/Group | Armodafinil
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From Screening through end of treatment; median (full range) of treatment was 98 (5.0 to 326.0) days.
Arm/Group | Armodafinil
Serious Adverse Events (participants affected / at risk) | 1/47
Other Adverse Events (participants affected / at risk) | 29/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Armodafinil (N=47)
Psychotic Disorder (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Armodafinil (N=47)
Nausea (Gastrointestinal disorders) | 3
Dry mouth (Gastrointestinal disorders) | 2
Feeling jittery (General disorders) | 2
Upper respiratory tract infection (Infections and infestations) | 4
Muscle strain (Injury, poisoning and procedural complications) | 2
Weight decreased (Investigations) | 2
Muscle tightness (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 7
Insomnia (Psychiatric disorders) | 3
Anxiety (Psychiatric disorders) | 2

LIMITATIONS AND CAVEATS:
The sponsor's decision to terminate the study early resulted in the small number of study participants, and related limitations to the interpretation of the study results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.